CLINICAL TRIAL: NCT05664919
Title: Safety and Effectiveness of SA58 Nasal Spray Against COVID-19 Infection in Medical Personnel：An Open-label, Blank-controlled Study
Brief Title: Efficacy and Safety of Anti-COVID-19 Antibody SA58 Nasal Spray to Prevent Infection in High-risk Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-SA58-0001
Record Dates: First submitted 2022-12-23; First posted 2022-12-27 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug group (Experimental): 3500 participants will use SA58 Nasal Spray in drug group.
  Interventions: Drug: SA58 Nasal Spray
- Blank control group (No Intervention): 3500 participants won't be given medication in blank control group.

INTERVENTIONS:
Drug: SA58 Nasal Spray — SA58 nasal spray , provided by Sinovac Life Sciences Co. , Ltd. mainly consists of neutralizing antibody of COVID-19, with 5 mg neutralizing antibody of COVID-19 per ml, 20 sprays per bottle.
  Arms: Drug group

SUMMARY:
This is an open, blank controlled clinical trial to evaluate the efficacy and safety of SA58 nasal spray in the prevention COVID-19 infection among health care workers at high risk of SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This is an open, blank controlled clinical trial to evaluate the efficacy and safety of SA58 nasal spray in the prevention COVID-19 infection among health care workers at high risk of SARS-CoV-2 infection.The investigational drug was manufactured by Sinovac Life Sciences Co. , Ltd.A total of 7000 medical personnel will be involved in this study: 3500 will use SA58 Nasal Spray in the drug group, and 3500 not use SA58 Nasal Spray in the blank control group. The medication is self-administered intranasally 1~2 times per day with an interval of 6 hours for about 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Medical staff working in the designated COVID-19 hospitals and Fangcang shelter hospitals (alternate care sites) of COVID-19 cases in Hohhot;
* Subjects were 18 years of age and older and in good health;
* Subjects volunteered to use COVID-19 neutralizing antibody nasal spray.

Exclusion Criteria:

* Previous history of severe allergies or sensitivity to inhaled allergens;
* Women were pregnant or breastfeeding;
* Subjects were unable to cooperate with nasal spray inhalation;
* Other conditions for which medication was not appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 infection rates | Up to 30 days(during case surveillance period)
  COVID-19 infection rates confirmed by RT-PCR among health care workers during the study period.

SECONDARY OUTCOMES:
Infection rates of asymptomatic and symptomatic COVID-19 patients | Up to 30 days(during case surveillance period)
  Infection rates of asymptomatic and symptomatic COVID-19 patients (i.e., confirmed cases) confirmed by RT-PCR during the study period.
Incidence of mild, normal, severe, and critical COVID-19 cases | Up to 30 days(during case surveillance period)
  Incidence of mild, normal, severe, and critical COVID-19 cases confirmed by RT-PCR during the study period.
The peak Ct value | Up to 30 days(during case surveillance period)
  The peak of Ct during the period of COVID-19 infection during the study period.
Differences in the number of days of negative RT-PCR | Up to 30 days(during case surveillance period)
  Differences in the number of days of negative RT-PCR during the period of COVID-19 infection during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Zhang, Principal Investigator — Inner Mongolia Fourth Hospital
Locations (1):
- Inner Mongolia Fourth Hospital, Hohhot, The Inner Mongolia Autonomous Region, China